CLINICAL TRIAL: NCT05437796
Title: Using the Immersive Virtual Reality for the Management of Anxiety and Pain in Orthopedic Surgery
Brief Title: Immersive Virtual Reality in Orthopedics
Acronym: IVR-Ortho
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Montauban (Other)
Responsible Party: Principal Investigator, Edmundo PEREIRA DE SOUZA NETO, Principal Investigator, Centre Hospitalier de Montauban
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A00005-34
Record Dates: First submitted 2022-06-19; First posted 2022-06-29 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Virtual Reality; Orthopedic
Keywords: Anxiety; Immersive virtual reality; Orthopedics; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to evaluate the effectiveness of hypnotic virtual reality support on the patient's state of anxiety before and after prosthetic knee surgeries under spinal anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnotic virtual reality support (Active Comparator): Hypnotic virtual reality support using hypnosis software Hypno-VR® (Strasbourg, France) paired with VR headsets Oculus VR® (Menlo Park, CA, USA)
  Interventions: Device: Hypnotic virtual reality support using hypnosis software Hypno-VR®
- Without hypnotic virtual reality support (Sham Comparator)
  Interventions: Device: No Hypnotic virtual reality

INTERVENTIONS:
Device: Hypnotic virtual reality support using hypnosis software Hypno-VR® — Hypnosis software Hypno-VR® (Strasbourg, France) paired with VR headsets Oculus VR® (Menlo Park, CA, USA)
  Other Names: Hypnotic virtual reality
  Arms: Hypnotic virtual reality support
Device: No Hypnotic virtual reality — Group without Hypnotic virtual reality
  Arms: Without hypnotic virtual reality support

SUMMARY:
Interventions may be a particular source of anxiety for some patients, and the management of surgical pain is still a real challenge. In order to avoid the side effects of medications, a lot of caregivers are turning to complementary medicines.

The prosthetic knee surgeries are painful and anxiety-provoking acts. At the hospital of Montauban, to relieve patients' pain, we offer them a therapeutic regimen with regional anesthesia (spinal anesthesia). We also use accompaniment hypnotic virtual reality to the management of anxiety and pain patients.

DETAILED DESCRIPTION:
Interventions may be a particular source of anxiety for some patients, and the management of surgical pain is still a real challenge. In order to avoid the side effects of medications, a lot of caregivers are turning to complementary medicines.

The prosthetic knee surgeries are painful and anxiety-provoking acts. At the hospital of Montauban, to relieve patients' pain, we offer them a therapeutic regimen with regional anesthesia (spinal anesthesia). We also use accompaniment hypnotic virtual reality to the management of anxiety and pain patients.

Despite a high level of approval of patients (according our satisfaction surveys) concerning hypnotic virtual reality, we want to evaluate our practice. Thus, in the future, we can invest in this type of material and make it available to a larger number of patients, but only if complementary care proves its effectiveness.

The purpose of this study is to evaluate the effectiveness of hypnotic virtual reality support on the patient's state of anxiety before and after prosthetic knee surgeries under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients for prosthetic knee surgery under spinal anesthesia
* Patient who has received appropriate information and has provided informed consent
* Patient with French social security system

Exclusion Criteria:

* Patient under general anaesthesia
* Patients treated in conventional inpatient care or in the traditional ambulatory circuit
* Patient under guardianship or trusteeship
* Minor patient < 18 years of age
* Patient who has not provided informed consent or who cannot submit to the study protocol
* Patient suffering from cognitive disorders (ex: Alzheimer's disease)
* Patients who are deaf or hearing-impaired or epilepsy
* Infected patient or identified as carrier of an infectious agent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-10-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of state of anxiety Spielberger | 60 minutes
  Questionnaire state of anxiety Spielberger: The Anxiety-State Scale assesses the feelings of apprehension, tension, nervousness and anxiety that the subject feels anxiety when the situation.
  The total score ranges from 20 - 80. The following guidelines are recommended for the interpretation of scores:
  Minus than 35 normal or no anxiety; 36 to 45, mild anxiety; 46 to 55, moderate anxiety; 56 to 65 severe anxiety; more than 65 severe anxiety.
Measurement of general anxiety Spielberger | 60 minutes
  Questionnaire general anxiety Spielberger: This questionnaire assesses your anxiety in life in general, and refers to trait anxiety. It is a stable disposition of personality.
  The total score ranges from 20 - 80. The following guidelines are recommended for the interpretation of scores:
  Minus than 35 normal or no anxiety; 36 to 45, mild anxiety; 46 to 55, moderate anxiety; 56 to 65 severe anxiety; more than 65 severe anxiety.

SECONDARY OUTCOMES:
Effectiveness of hypnotic virtual reality: | 48 hours
  The secondary objective of this research is to evaluate the effectiveness of hypnotic virtual reality:
  * On pain using evaluation visual analog scale (VAS) pain, graduated from 0 to 10, measured in the first 48 hours after surgery
  * On patient satisfaction using the Likert scale. The Likert scale is very popular and is often used in marketing research. It makes it possible to have nuances in the answers of respondents. Unlike scales dichotomous (yes / no), it makes it possible to have different degrees of judgment in analyzing the results. According to Likert, the most reliable measurement scales are those in seven ways:
    * Not at all satisfied
    * Unsatisfied
    * Somewhat dissatisfied
    * Neutral
    * Rather satisfied
    * Satisfied
    * Very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Edmundo Pereira de Souza Neto, Montauban, Tarn Et Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Askay SW, Patterson DR, Sharar SR. VIRTUAL REALITY HYPNOSIS. Contemp Hypn. 2009 Mar;26(1):40-47. doi: 10.1002/ch.371. PMID 20737029
- [Background] Benhaiem JM, Attal N, Chauvin M, Brasseur L, Bouhassira D. Local and remote effects of hypnotic suggestions of analgesia. Pain. 2001 Jan;89(2-3):167-73. doi: 10.1016/s0304-3959(00)00359-6. PMID 11166472
- [Background] Sharar SR, Miller W, Teeley A, Soltani M, Hoffman HG, Jensen MP, Patterson DR. Applications of virtual reality for pain management in burn-injured patients. Expert Rev Neurother. 2008 Nov;8(11):1667-74. doi: 10.1586/14737175.8.11.1667. PMID 18986237
- [Background] Hoffman HG, Patterson DR, Soltani M, Teeley A, Miller W, Sharar SR. Virtual reality pain control during physical therapy range of motion exercises for a patient with multiple blunt force trauma injuries. Cyberpsychol Behav. 2009 Feb;12(1):47-9. doi: 10.1089/cpb.2008.0056. PMID 19018695
- [Background] Borteyrou X, Bruchon-Schweitzer M, Spielberger CD. [The French adaptation of the STAXI-2, C.D. Spielberger's State-trait anger expression inventory]. Encephale. 2008 Jun;34(3):249-55. doi: 10.1016/j.encep.2007.06.001. Epub 2007 Oct 10. French. PMID 18558145
- [Background] Spielberger CD, Auerbach SM, Wadsworth AP, Dunn TM, Taulbee ES. Emotional reactions to surgery. J Consult Clin Psychol. 1973 Feb;40(1):33-8. doi: 10.1037/h0033982. No abstract available. PMID 4688678
- [Background] Hodgues WF, Spielberger CD. An indicant of trait or state anxiety? J Consult Clin Psychol. 1969 Aug;33(4):430-4. doi: 10.1037/h0027813. No abstract available. PMID 5810587
- [Background] Williamson A. What is hypnosis and how might it work? Palliat Care. 2019 Jan 31;12:1178224219826581. doi: 10.1177/1178224219826581. eCollection 2019. No abstract available. PMID 30728719
- [Background] Ahmadpour N, Randall H, Choksi H, Gao A, Vaughan C, Poronnik P. Virtual Reality interventions for acute and chronic pain management. Int J Biochem Cell Biol. 2019 Sep;114:105568. doi: 10.1016/j.biocel.2019.105568. Epub 2019 Jul 12. PMID 31306747
- [Background] Chan E, Hovenden M, Ramage E, Ling N, Pham JH, Rahim A, Lam C, Liu L, Foster S, Sambell R, Jeyachanthiran K, Crock C, Stock A, Hopper SM, Cohen S, Davidson A, Plummer K, Mills E, Craig SS, Deng G, Leong P. Virtual Reality for Pediatric Needle Procedural Pain: Two Randomized Clinical Trials. J Pediatr. 2019 Jun;209:160-167.e4. doi: 10.1016/j.jpeds.2019.02.034. Epub 2019 Apr 29. PMID 31047650
- [Background] Spiegel B, Fuller G, Lopez M, Dupuy T, Noah B, Howard A, Albert M, Tashjian V, Lam R, Ahn J, Dailey F, Rosen BT, Vrahas M, Little M, Garlich J, Dzubur E, IsHak W, Danovitch I. Virtual reality for management of pain in hospitalized patients: A randomized comparative effectiveness trial. PLoS One. 2019 Aug 14;14(8):e0219115. doi: 10.1371/journal.pone.0219115. eCollection 2019. PMID 31412029
- [Background] Carl E, Stein AT, Levihn-Coon A, Pogue JR, Rothbaum B, Emmelkamp P, Asmundson GJG, Carlbring P, Powers MB. Virtual reality exposure therapy for anxiety and related disorders: A meta-analysis of randomized controlled trials. J Anxiety Disord. 2019 Jan;61:27-36. doi: 10.1016/j.janxdis.2018.08.003. Epub 2018 Aug 10. PMID 30287083
- [Background] Bani Mohammad E, Ahmad M. Virtual reality as a distraction technique for pain and anxiety among patients with breast cancer: A randomized control trial. Palliat Support Care. 2019 Feb;17(1):29-34. doi: 10.1017/S1478951518000639. Epub 2018 Sep 10. PMID 30198451
- [Background] Smith V, Warty RR, Sursas JA, Payne O, Nair A, Krishnan S, da Silva Costa F, Wallace EM, Vollenhoven B. The Effectiveness of Virtual Reality in Managing Acute Pain and Anxiety for Medical Inpatients: Systematic Review. J Med Internet Res. 2020 Nov 2;22(11):e17980. doi: 10.2196/17980. PMID 33136055
- [Background] Anderson PL, Molloy A. Maximizing the impact of virtual reality exposure therapy for anxiety disorders. Curr Opin Psychol. 2020 Dec;36:153-157. doi: 10.1016/j.copsyc.2020.10.001. Epub 2020 Oct 15. PMID 33176268
- [Background] Gumaa M, Rehan Youssef A. Is Virtual Reality Effective in Orthopedic Rehabilitation? A Systematic Review and Meta-Analysis. Phys Ther. 2019 Oct 28;99(10):1304-1325. doi: 10.1093/ptj/pzz093. PMID 31343702
- [Background] Negrillo-Cardenas J, Jimenez-Perez JR, Feito FR. The role of virtual and augmented reality in orthopedic trauma surgery: From diagnosis to rehabilitation. Comput Methods Programs Biomed. 2020 Jul;191:105407. doi: 10.1016/j.cmpb.2020.105407. Epub 2020 Feb 21. PMID 32120088